CLINICAL TRIAL: NCT06856772
Title: Randomized Comparison of Morning Versus Bedtime Administration of Statins: A Cardiovascular Circadian Chronotherapy (C3) Trial
Acronym: STATIN-C3
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Tor Biering-Sørensen (Other)
Collaborators: Herlev and Gentofte Hospital (Other)
Responsible Party: Sponsor-Investigator, Tor Biering-Sørensen, MD, PhD, MPH, Herlev and Gentofte Hospital
Organization: Herlev and Gentofte Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: STATIN-C3
Record Dates: First submitted 2025-02-20; First posted 2025-03-04 (Actual); Last update posted 2025-03-04 (Actual); Status verified 2025-02

CONDITIONS: Cardiovascular Diseases (CVD); Drug Effect; Atherosclerosis Cardiovascular Disease
Keywords: Statin; Circadian Rhythm; Randomized Controlled Trial; Pragmatic; Outcomes; Cardiovascular disease; Prevention
MeSH Terms: conditions — Cardiovascular Diseases | interventions — Hydroxymethylglutaryl-CoA Reductase Inhibitors; Simvastatin; Atorvastatin; Rosuvastatin Calcium; Pravastatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Statin at bedtime (Experimental): Statin in the current prescribed dose
  Interventions: Drug: Statin in the evening (such as Simvastatin, Atorvastatin, Rosuvastatin, Pravastatin)
- Statin in the morning (Experimental): Statin in the current prescribed dose
  Interventions: Drug: Statin in the morning (such as Simvastatin, Atorvastatin, Rosuvastatin, Pravastatin)

INTERVENTIONS:
Drug: Statin in the evening (such as Simvastatin, Atorvastatin, Rosuvastatin, Pravastatin) — Participants will be instructed to take their Statin daily at approx. 8PM-12AM.
  Arms: Statin at bedtime
Drug: Statin in the morning (such as Simvastatin, Atorvastatin, Rosuvastatin, Pravastatin) — Participants will be instructed to take their statin upon awakening/or with their breakfast (approx. 6AM-10AM).
  Arms: Statin in the morning

SUMMARY:
Statins inhibit hydroxy-methylglutaryl coenzyme A (HMG-CoA) reductase which catalyzes the rate-limiting step in cholesterol synthesis. This in turn leads to reductions in concentrations of low-density lipoprotein (LDL) cholesterol and C-reactive protein which reduces the risk of incident atherosclerotic events among individuals both with and without a history of atherosclerotic cardiovascular Several pilot studies have suggested potential benefits of taking statin in the evening rather than in the morning.

The primary objective of this study is to examine whether statin administration at bedtime versus in the morning provides a superior reduction in the incidence of major adverse cardiovascular events among patients with or without established atherosclerotic cardiovascular disease, who are already taking statin.

DETAILED DESCRIPTION:
The study is a pragmatic, registry-based, open-label, randomized controlled trial combining the utilization of the Danish nationwide health registries and the official Danish electronic letter system (Digital Post/eBoks) into an innovative, decentralized trial requiring no study visits from participants. The nationwide health registries will be used for identification of potential participants and data collection, including baseline information and follow-up data, while the electronic letter system will be used for sending recruitment letters and communicating with participants. Study participants will provide electronic informed consent from home before inclusion and randomization.

The trial will include patients currently in statin treatment regardless of the presence or absence of established cardiovascular disease. Participants will be randomized 1:1 to either statin administration at bedtime or in the morning. The trial is event-driven.

ELIGIBILITY:
Inclusion Criteria:

* Age >=18 years
* Current treatment with atorvastatin 10-80 mg, rosuvastatin 5-40 mg, simvastatin 10-80 mg or pravastatin 20-40 mg (as recorded in the Danish National Prescription Registry and confirmed by the participant via questionnaire)
* Signed informed consent

Exclusion Criteria:

* none

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42000 (Estimated)
Dates: Start 2025-02-28 (Estimated); Primary Completion 2028-03-28 (Estimated); Study Completion 2028-03-28 (Estimated)

PRIMARY OUTCOMES:
Composite of hospitalization for myocardial infarction, hospitalization for stroke or cardiovascular death | Will be assessed in a time-to-first-event approach from date of randomization until end of study (up til 5 years).
  For Hospitalizations: Inpatient, at least 1 night

SECONDARY OUTCOMES:
Hospitalization for myocardial infarction | Will be assessed in a time-to-first-event approach from date of randomization until end of study (up til 5 years).
  Inpatient, at least 1 night
Hospitalization for stroke | Will be assessed in a time-to-first-event approach from date of randomization until end of study (up til 5 years).
  Inpatient, at least 1 night
Cardiovascular death | Will be assessed in a time-to-first-event approach from date of randomization until end of study (up til 5 years).
All-cause death | Will be assessed in a time-to-first-event approach from date of randomization until end of study (up til 5 years).

OTHER OUTCOMES:
Hospitalization for unstable angina | Will be assessed in a time-to-first-event approach from date of randomization until end of study (up til 5 years).
  Inpatient, at least 1 night
Coronary revascularization | Will be assessed in a time-to-first-event approach from date of randomization until end of study (up til 5 years).
Any arterial revascularization | Will be assessed in a time-to-first-event approach from date of randomization until end of study (up til 5 years).
Any venous thromboembolism | Will be assessed in a time-to-first-event approach from date of randomization until end of study (up til 5 years).
  The incidence of Any venous thromboembolism
Hospitalization for heart failure | Will be assessed in a time-to-first-event approach from date of randomization until end of study (up til 5 years).
  The incidence of Hospitalization for heartfailure. For hospitalizations: Inpatient, at least 1 night
Hospitalization for rhabdomyolysis | From date of randomization until end of study (up til 5 years)
  The incidence of Hospitalization for rhabdomyolysis, Inpatient, at least 1 night.
Any incident cancer | From date of randomization until end of study (up til 5 years)
  The incidence of any cancer
Any incident renal disorder | From date of randomization until end of study (up til 5 years)
  The incidence of any renal disorder
Any incident hepatic disorder | From date of randomization until end of study (up til 5 years)
  The incidence of any hepatic disorder
Bleeding episodes requiring hospitalization | From date of randomization until end of study (up til 5 years)
  The incidence of any bleeding episodes requiring hospitalization. For hospitalizations: Inpatient, at least 1 night.
Any Incident Diabetes mellitus | From date of randomization until end of study (up til 5 years)
  The incidence of diabetes mellitus
Plasma Lipid levels | From date of randomization until end of study (up til 5 years)
Plasma C-reactive protein level | From date of randomization until end of study (up til 5 years)
Time of day of hospitalization for myocardial infarction | From date of randomization until end of study (up til 5 years)
  The time of hospitalization will be expressed as the hour of the beginning of the hospitalization
Time of day of hospitalization for stroke | From date of randomization until end of study (up til 5 years)
  The time of hospitalization will expressed as the hour of the beginning of the hospitalization.

CONTACTS AND LOCATIONS:
Locations (1):
- Center for Translational Cardiology and Pragmatic Randomized Trials, Department of Cardiology, Copenhagen University Hospital - Herlev and Gentofte, Hellerup, Denmark

IPD SHARING:
Plan to Share IPD: Yes
Baseline and endpoint data will be collected from Danish administrative health registries, which are subject to Danish legislation and can only be made available to a third party under certain conditions. Please contact the sponsor in case of any inquiries.